CLINICAL TRIAL: NCT01340872
Title: A Prospective, Multicentre, Randomised, Double-blind, Placebo Controlled Study With Oral ST10-021 for the Treatment of Iron Deficiency Anaemia in Subjects With Quiescent Ulcerative Colitis Where Oral Ferrous Preparations Have Failed or Cannot be Used (AEGIS 1)
Brief Title: Safety and Efficacy Study of Oral Ferric Iron To Treat Iron Deficiency Anaemia in Quiescent Ulcerative Colitis (AEGIS-1)
Acronym: AEGIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST10-01-301; 2010-023588-16 (EudraCT Number)
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Iron Deficiency Anaemia; Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: iron deficiency; anaemia; inflammatory bowel disease; ulcerative colitis
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases; Colitis, Ulcerative; Iron Deficiencies; Anemia | interventions — ferric trimaltol; ferric maltol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ST10 (Experimental): ST10 (Ferric Maltol) 30mg capsules, taken orally twice a day
  Interventions: Drug: ST10-021
- Placebo (Placebo Comparator): Matching placebo capsules for ST10 (Ferric Maltol), taken orally twice a day
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: ST10-021 — 30 mg capsules to be taken orally twice a day for 12 weeks
  Other Names: Ferric Trimaltol; Ferric maltol; Feraccru
  Arms: ST10
Drug: Placebo Comparator — Matching sugar pill to be taken orally twice a day for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether ST10-021, an oral ferric iron preparation, is safe and effective in the treatment of iron deficiency anaemia (IDA) in subjects with non-active ulcerative colitis (UC).

DETAILED DESCRIPTION:
As no curative treatment is currently available for ulcerative colitis (UC), treatment options are restricted to controlling symptoms, maintaining remission and preventing relapse. As such, treatment of iron deficiency anaemia (IDA), a key symptom of the disease, is integral to the medical management of UC. Iron deficiency anaemia in UC is a chronically debilitating disorder which has a significant impact on the quality of life of affected subjects. Characteristic symptoms of IDA include chronic fatigue, headache, and subtle impairment of cognitive function. Up to one third of subjects with UC suffer from recurrent anaemia, with hospitalization required in severe cases. First line standard therapy for mild to moderate IDA in UC is typically oral ferrous products (OFP), however this is often not successful. Many subjects are intolerant and suffer from continuously occurring side effects, occasional exacerbation of inflammatory lesions and failure to correct iron deficiency. Common adverse effects of OFP include nausea, epigastric discomfort and constipation, all of which are dose-related and appear especially evident in subjects with UC.

As compared to oral ferrous iron, oral ferric iron can be administered with improved tolerability and the total dose exposure of unabsorbed iron within the gastrointestinal tract is significantly reduced. In addition, the iron is retained in its chelated form if not absorbed and this may reduce the risk of irritation within the gastrointestinal tract. Clinical studies conducted to date provide preliminary evidence for the therapeutic potential of ST10-021 in patients with IDA in Inflammatory Bowel Disease, including UC.

The purpose of this study is to determine whether ST10-021 is safe and effective in the treatment of IDA in subjects with non-active UC. In an effort to target an underserved population, the study will include only those subjects who have failed OFP in the past, or where OFP cannot be used.

ELIGIBILITY:
Inclusion Criteria:

* Competency to understand and sign the IEC/IRB approved informed consent form prior to any study mandated procedure, and willing/able to comply with study requirements
* Age ≥ 18 years
* Current diagnosis of quiescent UC as defined by SCCAI score of < 4
* Current diagnosis of IDA as defined by Hb ≥ 9.5 g/dl and <12.0 g/dl for women and ≥ 9.5 g/dl and <13.0 g/dl for men; ferritin < 30 µg/l
* Prior OFP failure as defined per protocol
* If receiving protocol-allowed immunosuppressant must be on stable dose
* Females of childbearing potential must agree to use a reliable method of contraception

Exclusion Criteria:

* Anaemia due to any cause other than iron deficiency
* Intramuscular or intravenous injection or administration of depot iron preparation, blood infusions, or erythropoietin within 3 months
* Oral iron supplementation use within 1 month
* Use of immunosuppressant with known effect of anaemia induction within 1 month
* Vitamin B12 or Folic Acid injection/infusion within 4 weeks
* Untreated Vitamin B-12 or Folic Acid deficiency
* Known hypersensitivity or allergy to ST10-021 or components of the study medication, or contraindication for treatment with iron preparations
* Other chronic or acute inflammatory or infectious diseases
* Creatinine > 2.0 mg/dl
* AST or ALT levels ≥ 5 times the upper limit of normal
* Cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that may adversely affect the safety of the subject and/or efficacy of the study drug or severely limit the lifespan of the subject
* History of malignancy within the past 5 years (except in situ removal of basal cell carcinoma)
* Significant neurologic or psychiatric symptoms resulting in disorientation, memory impairment, or inability to report accurately that might interfere with treatment compliance, study conduct or interpretation of the results
* Participation in another interventional clinical study within 30 days or during the study
* Inmates of a psychiatric ward, prison, or other state institution
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Scheduled or expected hospitalization and/or surgery during the course of the study
* Females who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mallard, PhD, Study Director — Shield Therapeutics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gasche C, Ahmad T, Tulassay Z, Baumgart DC, Bokemeyer B, Buning C, Howaldt S, Stallmach A; AEGIS Study Group. Ferric maltol is effective in correcting iron deficiency anemia in patients with inflammatory bowel disease: results from a phase-3 clinical trial program. Inflamm Bowel Dis. 2015 Mar;21(3):579-88. doi: 10.1097/MIB.0000000000000314. PMID 25545376
- [Result] Schmidt C, Ahmad T, Tulassay Z, Baumgart DC, Bokemeyer B, Howaldt S, Stallmach A, Buning C; AEGIS Study Group. Ferric maltol therapy for iron deficiency anaemia in patients with inflammatory bowel disease: long-term extension data from a Phase 3 study. Aliment Pharmacol Ther. 2016 Aug;44(3):259-70. doi: 10.1111/apt.13665. Epub 2016 May 29. PMID 27237709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were selected from the general population attending each centre in UK, DE, AT or HU for routine care of their IBD and anaemia. Individuals interested in participating were invited for the Screening visit in order to assess eligibility. Written informed consent was obtained prior to conducting any study specific assessments.
Pre-assignment Details: Subjects were males or females aged ≥18 years with a confirmed diagnosis of UC, required to be in remission have a mild-to-moderate UC (defined by SCCAI score <4 at entry); mild-to-moderate IDA (Hb concentration ≥9.5 g/dL and <12.0 g/dL for females and ≥9.5 g/dL and <13.0 g/dL for males; serum ferritin levels <30 μg/L at Screening.
Groups:
- ST10: 30mg ST10 capsules BD - double-blind phase
- Placebo: Matching placebo for ST10 capsules - double-blind phase
- ST10 - Open-label Continuation From Active Arm in Double-blind: Open-label extension of ST10 active treatment arm from double-blind phase
- Placebo Switch to Open-label Extension ST10 Treatment: Open-label extension ST10 treatment arm for placebo subjects completing double-blind phase
Period: Double-blind Phase
Arm/Group | ST10 | Placebo | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Started | 64 | 64 | 0 (Not Applicable to double-blind phase) | 0 (Not Applicable to double-blind phase)
Completed | 55 | 53 | 0 (Not Applicable to double-blind phase) | 0 (Not Applicable to double-blind phase)
Not Completed | 9 | 11 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Open-label Phase
Arm/Group | ST10 | Placebo | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Started | 0 (Not Applicable to open-label phase) | 0 (Not Applicable to open-label phase) | 50 (Only subjects in DE, UK and HU could enter the open-label extension (OLE); OLE rejected by EC in AT) | 47 (Only subjects in DE, UK and HU could enter the open-label extension (OLE); OLE rejected by EC in AT)
Completed | 0 (Not Applicable to open-label phase) | 0 (Not Applicable to open-label phase) | 37 | 36
Not Completed | 0 | 0 | 13 | 11
Not completed — Physician Decision | 0 | 0 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 8 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 6
Not completed — Worsening of IBD | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Potential subjects were screened for eligibility to participate based on their demographics, medical/surgical history, physical examination, concomitant medications, vital signs, clinical laboratory tests (including pregnancy test for females of child-bearing potential) and current IBD disease status (based on SCCAI clinical score). FAS - Safety
Groups:
- ST10: ST10: 30 mg Ferric Maltol capsules taken orally twice a day during a 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
- Placebo: Matching Placebo capsules taken orally twice a day during a 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
- Total: Total of all reporting groups
Arm/Group | ST10 | Placebo | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 63 | 125
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.52) | 38.5 (12.3) | 39.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 24 | 21 | 45
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 10 | 25
  Hungary | 11 | 15 | 26
  Germany | 35 | 32 | 67
  Austria | 4 | 6 | 10
Duration of ulcerative colitis (years) [Mean (Standard Deviation); unit: years] — Duration of ulcerative colitis (years); for participants with UC
  years | 9.0 (8.28) | 10.99 (11.43) | 9.99 (9.8)
Time since last IBD flare-up (months) [Mean (Standard Deviation); unit: months] — Time since last IBD flare-up (months) recorded at baseline
  months | 24.8 (59.16) | 21.51 (38.46) | 23.2 (48.4)
Time since last OFP dose (months) [Mean (Standard Deviation); unit: months] — Time since last prior oral ferrous product (OFP) dose (months)
  months | 36.17 (40.1) | 33.34 (44.04) | 34.76 (41.7)
Haemoglobin concentration at baseline [Mean (Standard Deviation); unit: g/dL] — Haemoglobin concentration at baseline of the 12 week double-blind phase
  g/dL | 11 (1.03) | 11.1 (0.85) | 11.05 (0.93)
Serum Ferritin concentration at baseline [Mean (Standard Deviation); unit: μg/L] — Serum Ferritin concentration at baseline of the 12 week double-blind phase
  μg/L | 8.6 (6.8) | 8.2 (6.5) | 8.4 (6.6)
TSAT% at baseline [Mean (Standard Deviation); unit: percentage] — TSAT% (transferrin saturation %) at baseline of the 12 week double-blind phase
  percentage | 10.6 (11.7) | 9.5 (7.5) | 10.05 (9.6)
Irritable Bowel Disease Questionnaire (IBDQ) score at baseline [Mean (Standard Deviation); unit: score on a scale] — Irritable Bowel Disease Questionnaire (IBDQ) score at baseline (randomisation) of the 12 week double-blind phase.
  The IBDQ was developed as an activity index for determining the effect of Ulcerative Colitis symptoms on perceived quality of life. It is a 32-item questionnaire with four dimensions: bowel function, emotional status, systemic symptoms and social function. Total IBDQ score ranges from 32 to 224, with higher scores indicating better quality of life. The score of patients in remission usually is between 170 and 190.
  score on a scale | 175.0 (30.92) | 171.0 (33.56) | 173.02 (32.23)
Simple Clinical Colitis Activity Index (SCCAI) score at baseline [Mean (Full Range); unit: score on a scale] — Simple Clinical Colitis Activity Index (SCCAI) score at baseline (randomisation) of the 12-week double-blind phase (in participants with UC).
  The SCCAI is a diagnostic and research questionnaire used to assess the severity of symptoms in people who suffer from UC. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  The score is determined by asking the person with UC questions regarding:
  * bowel frequency at day/night
  * urgency of defecation
  * blood in stool
  * general health
  * extracolonic manifestations
  score on a scale | 1.8 [0 to 3] | 1.4 [0 to 3] | 1.6 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin (Hb) Concentration From Baseline to Week 12 (Full Analysis Set, FAS)
Description: Primary efficacy endpoint, defined as the change in Hb concentration from Baseline to Week 12. Baseline was defined as the pre-dose Hb concentration measured at the Randomisation Visit (Week 0). Missing Randomisation Hb values were replaced by Screening Hb values, if the randomisation was within the protocol-specified window. Hb concentration (g/dL) was analysed by a central laboratory from blood samples collected at every clinic visit: Screening, Randomisation (Week 0), Weeks 4, 8, 12, 14, 16, 20, 24, 36, 48, 64, Weeks 14 to 64 were open-label. The baseline, absolute concentration and change from baseline in Hb at all post-randomisation visits were listed and summarised by week using descriptive statistics. An analysis of covariance (ANCOVA) was used to analyse the primary endpoint; this included treatment, gender and disease as factors and baseline Hb as a covariate.
Time Frame: Baseline to Week 12 - double-blind phase
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- ST10: ST10: 30 mg Ferric Maltol capsules taken orally twice a day during 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
- Placebo: Matching Placebo capsules taken orally twice a day during 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 58 | 53
g/dL | 2.26 (1.184) | 0.01 (0.764)
Statistical Analysis 1: Comparison: ST10 vs Placebo; ANCOVA for primary endpoint, Change in Hb concentration from Baseline to Week 12 in double-blind phase, FAS; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.18, 97.5% CI 1-sided [lower limit 1.81], Standard Error of Mean 0.19

2. Secondary Outcome: Proportion of Subjects That Achieved ≥1 g/dL Change From Baseline in Hb Concentration at Week 12 (Full Analysis Set, FAS)
Description: Logistic regression analysis of proportion of subjects that achieved ≥1 g/dL change from baseline in Hb concentration at Week 12 in the double-blind phase
Time Frame: Subjects that achieved ≥1 g/dL change from baseline in Hb concentration at Week 12 - double-blind phase
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 64 | 64
Participants
  Yes | 50 | 7
  No | 14 | 57

3. Secondary Outcome: Proportion of Subjects That Achieved ≥2 g/dL Change From Baseline in Hb Concentration at Week 12 (Full Analysis Set, FAS)
Description: Logistic regression analysis of proportion of subjects that achieved ≥2 g/dL change from baseline in Hb concentration at Week 12 in the double-blind phase
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- ST10: ST10: 30 mg Ferric Maltol capsules taken orally twice a day during 12-week double-blind phase.
- Placebo: Matching Placebo capsules taken orally twice a day during 12-week double-blind phase.
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 64 | 64
Participants
  Yes | 36 | 0
  No | 28 | 64

4. Secondary Outcome: Proportion of Subjects That Achieved Hb Concentration Within Normal Range at Week 12 (Full Analysis Set, FAS)
Description: Logistic regression analysis of proportion of subjects that achieved Hb concentration within normal range at Week 12 - end of double-blind phase
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 64 | 64
Participants
  Yes | 42 | 8
  No | 22 | 56

5. Secondary Outcome: Change in Hb Concentration From Baseline to Week 4 (Full Analysis Set, FAS)
Description: ANCOVA analysis of the change in Hb concentration from Baseline to Week 4 of the double-blind phase - Full Analysis Set, multiple imputation
Time Frame: Baseline to Week 4 - double-blind phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 59 | 61
g/dL | 1.08 (0.676) | 0 (0.67)
Statistical Analysis 1: Comparison: ST10 vs Placebo; ANCOVA analysis of the change in Hb concentration from Baseline to Week 4 of the double-blind phase - Full Analysis Set, multiple imputation; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.04, 97.5% CI 1-sided [lower limit 0.82], Standard Error of Mean 0.11

6. Secondary Outcome: Change in Hb Concentration From Baseline to Week 8 (Full Analysis Set, FAS)
Description: ANCOVA analysis of Change in Hb concentration from Baseline to Week 8 of double-blind phase - FAS, multiple imputation
Time Frame: Baseline to Week 8 - double-blind phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 59 | 56
g/dL | 1.79 (1.037) | 0.04 (0.722)
Statistical Analysis 1: Comparison: ST10 vs Placebo; ANCOVA analysis of Change in Hb concentration from Baseline to Week 8 of double-blind phase - FAS, multiple imputation; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.73, 97.5% CI 1-sided [lower limit 1.43], Standard Error of Mean 0.15

7. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 16 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 16 (FAS), after 12-week double-blind phase and first 4 weeks of open-label ST10 treatment.
Time Frame: Baseline to Week 16 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 46 | 45
g/dL | 2.34 (1.281) | 1.04 (1.023)

8. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 20 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 20 (FAS), after 12-week double-blind phase and then 8 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 20 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 43 | 43
g/dL | 2.45 (1.213) | 1.46 (1.056)

9. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 24 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 24 (FAS), after 12-week double-blind phase and then 12 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 24 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 43 | 41
g/dL | 2.68 (1.127) | 1.87 (1.195)

10. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 36 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 36 (FAS), after 12-week double-blind phase and then 24 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 36 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 41 | 36
g/dL | 2.85 (1.227) | 2.17 (1.048)

11. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 48 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 48 (FAS), after 12-week double-blind phase and then 36 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 48 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 40 | 37
g/dL | 3.09 (1.339) | 2.0 (1.191)

12. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 64 (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 64 (FAS), after 12-week double-blind phase and then 52 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 64 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 35 | 36
g/dL | 3.07 (1.457) | 2.19 (1.605)

13. Secondary Outcome: Change in Haemoglobin Concentration From Baseline to Week 64 EOS (Full Analysis Set, FAS)
Description: Change in Haemoglobin Concentration from Baseline to Week 64 EOS (FAS) - Week 64 was re-categorised as Week 64 EOS for those subjects who withdrew from the study early and the 'Week 64' visit was outside the visit window of 64 weeks ± 2 days
Time Frame: Baseline to Week 64 EOS - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 10 | 17
g/dL | 1.32 (1.713) | 0.52 (1.417)

14. Secondary Outcome: Proportion of Subjects That Achieved Haemoglobin Concentration Within Normal Range at Week 16 (Full Analysis Set, FAS)
Description: Proportion of subjects that achieved Haemoglobin Concentration within normal range at Week 16 (Full Analysis Set), after 12-week double-blind phase and first 4 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 16 - open-label phase
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 46 | 45
Participants
  Yes | 36 | 17
  No | 10 | 28

15. Secondary Outcome: Proportion of Subjects That Achieved Haemoglobin Concentration Within Normal Range at Week 36 (Full Analysis Set, FAS)
Description: Proportion of subjects that achieved Haemoglobin Concentration within normal range at Week 36 (Full Analysis Set), after 12-week double-blind phase and 24 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 36 - open-label phase
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 41 | 36
Participants
  Yes | 35 | 29
  No | 6 | 7

16. Secondary Outcome: Proportion of Subjects That Achieved Haemoglobin Concentration Within Normal Range at Week 64 (Full Analysis Set, FAS)
Description: Proportion of subjects that achieved Haemoglobin Concentration within normal range at Week 64 (Full Analysis Set), after 12-week double-blind phase and 52 weeks of open-label ST10 treatment
Time Frame: Baseline to Week 64 - open-label phase
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 36 | 36
Participants
  Yes | 31 | 30
  No | 5 | 6

17. Other Pre Specified Outcome: Change in Haemoglobin Concentration From Baseline to Week 12 (Per Protocol Analysis Set, PPAS)
Description: ANCOVA sensitivity analysis of the Primary efficacy endpoint analysis on the PPAS - Change in Haemoglobin Concentration from Baseline to Week 12
Time Frame: Baseline to Week 12 - double-blind phase
Population: Per-Protocol Analysis Set - sensitivity analysis of primary endpoint
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 55 | 57
g/dL | 2.23 (0.13) | 0.05 (0.13)
Statistical Analysis 1: Comparison: ST10 vs Placebo; ANCOVA sensitivity analysis of the Primary efficacy endpoint analysis on the PPAS; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.18, 97.5% CI 1-sided [lower limit 1.87], Standard Error of Mean 0.17

18. Other Pre Specified Outcome: Change in Haemoglobin Concentration From Baseline to Week 12 (Full Analysis Set [FAS] LOCF)
Description: ANCOVA sensitivity analysis of the Primary efficacy endpoint analysis on the FAS LOCF - Change in Haemoglobin Concentration from Baseline to Week 12
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS LOCF - sensitivity analysis of primary endpoint
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 64 | 64
g/dL | 2.11 (0.12) | -0.03 (0.12)
Statistical Analysis 1: Comparison: ST10 vs Placebo; ANCOVA sensitivity analysis of the Primary efficacy endpoint analysis on the FAS LOCF - Change in Haemoglobin Concentration from Baseline to Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.15, 97.5% CI 1-sided [lower limit 1.82], Standard Error of Mean 0.16

19. Other Pre Specified Outcome: Change in Serum Ferritin Concentration From Baseline to Week 12 (Full Analysis Set, FAS)
Description: Change in serum Ferritin concentration from Baseline to Week 12 (Full Analysis Set), after 12-week double-blind phase
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 59 | 53
μg/dL | 17.3 (28.3) | 1.2 (7.85)

20. Other Pre Specified Outcome: Change in Serum Ferritin Concentration From Baseline to Week 64 (Full Analysis Set, FAS)
Description: Change in serum Ferritin concentration from Baseline to Week 64 (FAS), after 12-week double-blind phase and 52 weeks open-label ST10 treatment
Time Frame: Baseline to Week 64 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 36 | 36
μg/dL | 60.4 (93.35) | 36.6 (46.8)

21. Other Pre Specified Outcome: Change in Serum TSAT% From Baseline to Week 12 (Full Analysis Set, FAS)
Description: Change in serum TSAT% from Baseline to Week 12 (FAS), after 12-week double-blind phase
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS
Measure: Mean (Standard Deviation); unit: % serum TSAT
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 59 | 52
% serum TSAT | 18.0 (20.17) | -0.4 (7.82)

22. Other Pre Specified Outcome: Change in Serum TSAT% From Baseline to Week 64 (Full Analysis Set, FAS)
Description: Change in serum TSAT% from Baseline to Week 64 (Full Analysis Set), after 12-week double-blind phase and 52 weeks open-label ST10 treatment
Time Frame: Baseline to Week 64 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: % serum TSAT
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 36 | 36
% serum TSAT | 18.8 (12.46) | 17.7 (16.2)

23. Other Pre Specified Outcome: Irritable Bowel Disease Questionnaire (IBDQ) Score at Week 12 (Full Analysis Set, FAS)
Description: Irritable Bowel Disease Questionnaire (IBDQ) score at Week 12 (FAS), end of double-blind phase.
  The IBDQ was developed as an activity index for determining the effect of Ulcerative Colitis symptoms on perceived quality of life. It is a 32-item questionnaire with four dimensions: bowel function, emotional status, systemic symptoms and social function. Total IBDQ score ranges from 32 to 224, with higher scores indicating better quality of life. The score of patients in remission usually is between 170 and 190.
Time Frame: Week 12 - double-blind phase
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 60 | 60
score on a scale | 178.3 (32.36) | 176.3 (31.5)

24. Other Pre Specified Outcome: Irritable Bowel Disease Questionnaire (IBDQ) Score at Week 64 (Full Analysis Set, FAS)
Description: Irritable Bowel Disease Questionnaire (IBDQ) score at Week 64 (FAS), after 12-week double-blind phase and 52 weeks of open-label ST10 treatment.
  The IBDQ was developed as an activity index for determining the effect of Ulcerative Colitis symptoms on perceived quality of life. It is a 32-item questionnaire with four dimensions: bowel function, emotional status, systemic symptoms and social function. Total IBDQ score ranges from 32 to 224, with higher scores indicating better quality of life. The score of patients in remission usually is between 170 and 190.
Time Frame: Week 64 - open-label phase
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 37 | 36
score on a scale | 180.7 (30.14) | 177.2 (36.97)

25. Other Pre Specified Outcome: Change From Baseline in Simple Clinical Colitis Activity Index (SCCAI) Score at Week 12 (Full Analysis Set, FAS)
Description: Change from baseline in Simple Clinical Colitis Activity Index (SCCAI) score at Week 12 (FAS), end of double-blind phase (in subjects with UC).
  The SCCAI is a diagnostic and research questionnaire used to assess the severity of symptoms in people who suffer from UC. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  The score is determined by asking the person with UC questions regarding:
  * bowel frequency at day/night
  * urgency of defecation
  * blood in stool
  * general health
  * extracolonic manifestations
Time Frame: Baseline to Week 12 - double-blind phase
Population: FAS - participants with UC only
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ST10 | Placebo
Number analyzed (Participants) | 28 | 29
score on a scale | 0 [-2 to 5] | 0 [-1 to 5]

26. Other Pre Specified Outcome: Change From Baseline in Simple Clinical Colitis Activity Index (SCCAI) Score at Week 64 (Full Analysis Set)
Description: Change from baseline in Simple Clinical Colitis Activity Index (SCCAI) score at Week 64 (FAS), after 12-week double-blind phase and 52 weeks open-label ST10 treatment (in participants with UC only).
  The SCCAI is a diagnostic and research questionnaire used to assess the severity of symptoms in people who suffer from UC. The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
  The score is determined by asking the person with UC questions regarding:
  * bowel frequency at day/night
  * urgency of defecation
  * blood in stool
  * general health
  * extracolonic manifestations
Time Frame: Baseline to Week 64 - open-label phase
Population: FAS
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ST10 - Open-label Continuation From Active Arm in Double-blind | Placebo Switch to Open-label Extension ST10 Treatment
Number analyzed (Participants) | 19 | 19
score on a scale | 0 [-3 to 2] | 0 [-2 to 5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were solicited after informed consent and until 4 weeks after the last dose of study drug (at study completion or early termination).
Description: Subjects were expected to volunteer information about AEs they experienced. The Investigator/designee also questioned the subject at each visit about AEs and recorded these as well as all other AEs apparent. AEs/SAEs were monitored until they were resolved or determined to be due to a subject's on-going condition or inter-current illness.
Groups:
- ST10 - Safety Set, Double-blind Phase: Adverse events reported in the double-blind phase active treatment arm with ST10 (Ferric Maltol). ST10 30 mg capsules taken orally twice a day during a 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
- Placebo - Safety Set, Double-blind Phase: Adverse events reported in the double-blind phase placebo treatment arm. Matching placebo capsules for ST10 taken orally twice a day during a 12-week double-blind phase. For study participants in the UK, DE and HU only, the 12-week double-blind phase was followed by a 52-week open-label ST10 extension treatment phase.
- ST10 Continuation - Safety Set, Open-label Phase: Adverse events reported in the open-label extension phase for continuation of active treatment with ST10 (Ferric Maltol) from the double-blind phase active treatment arm.
- Placebo Switch to ST10 Treatment-Safety Set, Open-label Phase: Adverse events reported in the open-label extension phase from those subjects continuing treatment from the double-blind placebo arm; subjects commenced ST10 open-label treatment after completion of the double-blind phase at the Week 12 visit.
Arm/Group | ST10 - Safety Set, Double-blind Phase | Placebo - Safety Set, Double-blind Phase | ST10 Continuation - Safety Set, Open-label Phase | Placebo Switch to ST10 Treatment-Safety Set, Open-label Phase
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/64 | 8/50 | 2/47
Other Adverse Events (participants affected / at risk) | 39/64 | 46/64 | 40/50 | 35/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST10 - Safety Set, Double-blind Phase (N=64) | Placebo - Safety Set, Double-blind Phase (N=64) | ST10 Continuation - Safety Set, Open-label Phase (N=50) | Placebo Switch to ST10 Treatment-Safety Set, Open-label Phase (N=47)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesteatoma removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST10 - Safety Set, Double-blind Phase (N=64) | Placebo - Safety Set, Double-blind Phase (N=64) | ST10 Continuation - Safety Set, Open-label Phase (N=50) | Placebo Switch to ST10 Treatment-Safety Set, Open-label Phase (N=47)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (3)
Fatigue (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 5 (6) | 2 (2) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (7)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 4 (5) | 4 (4) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 8 (8) | 12 (14) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No